CLINICAL TRIAL: NCT06373666
Title: A Study to Evaluate the Adjustment Function of a Modified Spatz3 Adjustable Balloon (Spatz4).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spatz FGIA, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPZ4-02
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spatz4 Balloon (Experimental): Subject will be implanted with the Spatz4 gastric balloon for a period of up to 12 months. At 16 weeks an up adjustment will performed to evaluate the adjustment function.
  Interventions: Device: Spatz4 Adjustable Balloon System

INTERVENTIONS:
Device: Spatz4 Adjustable Balloon System — Implantation of Spatz4 Adjustable Balloon system for weight loss treatment for Overweight and Obese patients and Adjustment of the balloon volume at week 16

SUMMARY:
The purpose of this study is to evaluate the function of the adjustment procedure with the Spatz4 in subjects with a BMI ≥ 27.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the function of the adjustment procedure with the Spatz4 in subjects with a BMI ≥ 27.

Subjects will be studied in an open label study that will have one endpoint at 20 weeks. Up to 20 eligible subjects will undergo endoscopy and those without endoscopic contraindications will be implanted with the Spatz4 balloon. All subjects will follow a calorie restricted diet designed by the dietician. The initial diet will be liquid and will be advanced as per the dietician's recommendations. Changes in diet will depend on subject tolerance to the balloon and specific food intolerances and will be adjusted frequently by the dietician. The initial balloon volume will be 450 to 550 ml of 0.9% normal saline with 2 ml of a 1% solution of methylene blue. It is estimated, based on clinical studies, that approximately 10% of subjects will be intolerant in the first month and will require a down adjustment, wherein 150 ml of fluid will be removed from the balloon. An up adjustment will be performed at 16 weeks (±2 weeks) with the addition of 200-300 ml of 0.9% normal saline, as per section 1.7.2.1.3.3. The balloon adjustment procedure is done with an endoscopy procedure under the same sedation as the implantation procedure. The subjects will be followed for 2 weeks after the up-adjustment procedure, after which the study ends. Subjects will be given the option to continue the implantation period until 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI ≥ 27;
* Be male or female, between 18 and 65 years of age, inclusive;
* Have a history of excess weight (BMI ≥ 27 kg/m2) for at least 2 years and have failed more conservative weight-reduction alternatives, such as supervised diet, exercise and behavioral modification programs;
* Be willing to commit to a long-term low calorie (1000-1500 calories/day) supervised diet;
* Have reasonable weight loss expectations (accept a goal of losing up to 15% of body weight after 52 weeks);
* Be able to follow requirements outlined in the protocol, including complying with the visit schedule and behavioral modification program, and willing to undergo protocol-specific procedures, e.g., endoscopy, local sedation, general anesthesia, upper gastrointestinal radiography (UGI), electrocardiography (EKG), gastric motility testing, and/or clinical laboratory testing, and must be willing to take prescribed proton pump inhibitors (PPIs);
* Be able to provide written informed consent;
* Have successful completion of the pre-placement screening and educational programs supporting that the subject is an appropriate study candidate;
* Be willing to use contraception (e.g., birth control pills, condoms, abstinence) and avoid pregnancy during the study if female of child-bearing potential.

Exclusion Criteria:

* Previous history of esophageal, gastric or duodenal surgery, any bariatric surgery, any hiatal hernia surgery, bowel obstruction surgery, adhesive peritonitis, and/or hiatal hernia > 4 cm;
* A history of myocardial infarction in the previous 6 months: New York Heart Associate (NYHA) Class III or IV (heart failure) or cardiac arrhythmia (e.g. atrial fibrillation);
* History or symptoms of varices, bowel obstruction, congenital or acquired GI anomalies (e.g., atresias, stenosis, stricture, and/or diverticula), severe renal, hepatic, and/or pulmonary disease;
* History or symptoms of inflammatory bowel disease, such as Crohn's disease;
* History of unstable thyroid disease;
* History of uncontrolled gastro-esophageal reflux;
* Type I diabetes;
* History of dysphagia, esophageal stricture or esophageal food impaction;
* Poor general health, in the opinion of the Placing and/or Evaluating Investigator, or presence of a specific medical condition that would increase the risks associated with endoscopy and/or placement of the Spatz4;
* Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
* Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD);
* Specific diagnosed genetic or hormonal cause for obesity such as Prader Willi syndrome
* History or symptoms of esophageal or GI motility disorders (e.g., gastroparesis, achalasia, diffuse esophageal spasm) or symptoms of esophageal stricture;
* Ongoing treatment with anticoagulants, steroids, aspirin > 100 mg, non-steroidal anti-inflammatory drugs (NSAIDS), or other medications known to be gastric irritants, and inability or unwillingness to discontinue the use of these concomitant medications;
* Evidence of untreated psychiatric or eating disorders, such as major depression, schizophrenia, substance abuse;
* Pregnancy, breast-feeding, or intention of becoming pregnant during the study (if female of childbearing potential);
* A condition, or is in a situation, which in the Evaluating and/or Placing Investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Successful adjustment procedure at 16 ±2 weeks in > 85% of attempts. | 16 ± 2 weeks
  The study will have one endpoint: Proportion of subjects with successful adjustment procedure is greater than 85%

CONTACTS AND LOCATIONS:
Locations (1):
- Endohope Havířov s.r.o., Havířov, Czechia

IPD SHARING:
Plan to Share IPD: No